CLINICAL TRIAL: NCT01567540
Title: A Pilot Study to Evaluate the Clinical and Biological Tolerance of Sitagliptin With Pegylated Interferon alfa2a Plus Ribavirin Combination Therapy in Chronic Hepatitis C Patients
Brief Title: A Pilot Study Evaluating Safety of Sitagliptin Combined With Peg-IFN Alfa-2a + Ribavirin in Chronic Hepatitis C Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New treatments available, which prevents additional recruitment.
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10-54; 2011-000823-34 (EudraCT Number)
Record Dates: First submitted 2012-03-02; First posted 2012-03-30 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C; Interferon protein 10; Chemokine gradients; Sitagliptin
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DPPIV Inhibition (Experimental): The study includes an initial phase of 3 weeks with administration of sitagliptin (100 mg/d) as monotherapy, followed immediately by 12 weeks of triple therapy (sitagliptin 100 mg/d combined with peg-IFN alfa-2a and ribavirin).
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 100 mg Sitagliptin daily for 15 weeks

SUMMARY:
Hepatitis C infection is a major public health problem with nearly 175 million infected individuals worldwide. Although cure is possible, only 20-40% of patients spontaneously resolve infection and 40-80% of chronically infected patients (numbers vary depending on viral genotype) that receive pegylated-interferon-alfa2a/ribavirin therapy clear the virus and are sustained virologic responders (SVR). Still for many, the virus manages to circumvent natural immunity and current therapeutic strategies, resulting in significant morbidity and mortality.

To better define the distinct clinical outcomes of HCV infection many investigators have performed candidate molecules screens or transcriptional profiling in order to identify correlates of viral clearance. One molecule that has gained significant attention is CXCL10 (also known as interferon-gamma induced protein-10 or IP-10) as an important negative prognostic biomarker. Given that CXCL10 is produced by hepatocytes and mediates chemo-attraction of activated lymphocytes expressing the CXCL10-receptor, CXCR3, it is counter-intuitive as to why this chemokine correlates with therapeutic non-responsiveness.

The investigators hypothesized and have now demonstrated that CXCL10 is being cleaved in situ, resulting in the generation of an antagonist form of the chemokine. Based on the use of specific inhibitors, the investigators now propose to test whether protection of the agonist form of CXCL10 will increase responsiveness to peg-IFN-alfa2 / ribavirin therapy. This can be achieved using DPPIV inhibitors, targeting the enzyme responsible for N-terminal truncation of CXCL10. If safety is confirmed, the efficacy of DPPIV-inhibition in HCV patients will be tested in future trials that examine potential clearance benefits.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* For women, effective contraception during the trial and a negative pregnancy test (urine) before enrollment
* Patients naïve to prior hepatitis C treatment
* Confirmed HCV infection, based on the presence of HCV antibodies and plasma viremia allowing a measure of the circulating viral load
* Infection with HCV genotype 1 or 4
* Intent of treatment Alfa2 pegylated IFN-/ ribavirin

Exclusion Criteria:

* HBV Infection
* HIV Infection
* Severe anemia (Hb <7-8 g / dl)
* Renal failure (creatinine clearance <60 ml / min)
* Taking digoxin within 6 months of starting treatment.
* Taking immunosuppressants within 6 months of starting treatment
* History of serious hypersensitivity reaction (such as anaphylactic shock or angioedema) to sitagliptin
* Patients with type I and II diabetes
* Pregnancy or absence of effective contraception
* A person deprived of liberty by judicial or administrative decision
* Living conditions-suggesting an inability to track all scheduled visits by the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Safety (Number of adverse events, Toxicity grade > 3) | After Day 1 until the end of the trial, i.e. a duration of 15 weeks for each patient

SECONDARY OUTCOMES:
Change in Viral Load as compared to baseline | week 1, 2, 3 of sitagliptin monotherapy; week 2, 4, 12 of triple therapy
Metabolic studies: Oral glucose tolerance will be assessed | baseline, week 1 of sitagliptin monotherapy; week 2 of triple therapy
Immunologic study | baseline, week 1 and 3 of sitagliptin monotherapy; week 1, 2, 4, 12 of triple therapy
  Monitoring the short and long form of IP-10 as compared to the total plasma concentration (three distinct ELISA assays).
Immunologic study | baseline; week 1 and 3 of sitagliptin monotherapy; week 1, 2, 4, 12 of triple therapy
  Plasma concentration and activity of DPPIV (measured using an ELISA and a luciferase-based bioassay, respectively).
Immunologic study | baseline, week 1 and 3 of sitagliptin monotherapy; week 1, 2, 4, 12 of triple therapy.
  Frequency of CXCR3+ cells in circulation (monitored by FACS).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L. ALBERT, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (4):
- France (4):
  - Centre Hospitalier Victor Dupuy, Argenteuil
  - Centre Hospitalier Intercommunal Créteil, Créteil
  - Henri Mondor Hospital, Créteil
  - Cochin Hospital, Paris